CLINICAL TRIAL: NCT01533740
Title: Observational Study of the Impact of Circulating T Regulatory Cells (Tregs) on Clinical Outcome of Metastatic Colorectal Cancer (MCRC) Patients Treated With Standard Fluorouracil/Irinotecan/Bevacizumab First Line Therapy
Brief Title: Circulating Regulatory Lymphocytes and Outcome of Metastatic Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Vincenzo Formica, MD, PhD, University of Rome Tor Vergata
Other Study IDs: ONCOPTV-01-2012
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Bevacizumab; Irinotecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fluorouracil/irinotecan/levo-folinic acid/bevacizumab — standard first line chemotherapy with: bevacizumab 5 mg/kg intravenous (i.v.) infusion on day 1; irinotecan 180 mg/m2 i.v. infusion on day 1, levo-folinic acid 200 mg/m2 i.v. infusion on day 1, 5-fluorouracil 400 mg/m2 i.v. bolus on day 1 and 2,400 mg/m2 i.v. infusion over 46 hours; infusions repeated every 2 weeks
  Other Names: avastin (bevacizumab); campto (irinotecan)

SUMMARY:
Aim of the present study is to investigate whether baseline or early post-treatment (one month after treatment commencement) frequency of peripheral T regulatory lymphocytes (Tregs OR CD4+/CD25high/FOXP3+ T cells), known to suppress antitumor immune response, may influence long-term clinical outcome (i.e. radiological response, progression-free survival or overall survival) in metastatic colorectal cancer patients treated with a standard first-line chemotherapy including fluorouracil, irinotecan and bevacizumab

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically or cytologically confirmed diagnosis of metastatic colorectal cancer not amenable to surgery
* Adjuvant treatment ended ≥6 months before the study entry
* No prior exposure to irinotecan and/or bevacizumab in the adjuvant treatment
* No prior exposure to cytotoxic drugs for the metastatic disease
* At least one measurable lesion according to the RECIST criteria
* adequate laboratory parameters (Hemoglobin level ≥ 9.0 g/dL; Neutrophil count > 1.5 x 109/L; Platelets count >100 x 109/L; Total bilirubin <1.5 time the upper-normal limits (UNL) and ASAT (SGOT) and/or ALAT (SGPT) <2.5 x UNL, or <5 x UNL in case of liver metastases; alkaline phosphatase <2.5 x UNL, or <5 x UNL in case of liver metastases; PT-INR/PTT < 1.5 x UNL;Creatinine clearance > 50 mL/min or serum creatinine <1.5 x UNL; Urine dipstick of proteinuria < 2+)
* Written informed consent.
* Patients must be accessible for treatment and follow up.

Exclusion Criteria:

* Untreated brain metastases or spinal cord compression
* History of inflammatory bowel disease and/or acute or subacute bowel occlusion.
* Serious, non-healing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy.
* Uncontrolled hypertension.
* Clinically significant cardiovascular disease(cerebrovascular accidents ≤ 6 months, myocardial infarction ≤ 6 months, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication)
* Current or recent (within 10 days prior to study treatment start) ongoing treatment with anticoagulants for therapeutic purposes.
* Chronic, daily treatment with high-dose aspirin (>325 mg/day) or other medications known to predispose to gastrointestinal ulceration.
* Treatment with any investigational drug within 30 days prior to enrolment.
* Patients with known allergy to Chinese hamster ovary cell proteins, or any of the components of the study medications
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal and squamous cell carcinoma or cervical cancer in situ
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study.
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline
* Substance abuse, medical, psychological or social conditions that may interfere with the participation into the study or the evaluation of study results
* Patients unable to swallow oral medications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital setting, single-center study, metastatic colorectal cancer patients treated with standard first line chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Impact of Tregs frequency on overall survival | 12 months

SECONDARY OUTCOMES:
Impact of Tregs frequency progression free survival | 12 months
Impact of Tregs frequency radiologic response rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Formica, MD, PhD, Principal Investigator — 'Tor Vergata' University Hospital
Locations (1):
- 'Tor Vergata' University Hospital, Rome, Lazio, Italy

REFERENCES:
- [Derived] Formica V, Cereda V, di Bari MG, Grenga I, Tesauro M, Raffaele P, Ferroni P, Guadagni F, Roselli M. Peripheral CD45RO, PD-1, and TLR4 expression in metastatic colorectal cancer patients treated with bevacizumab, fluorouracil, and irinotecan (FOLFIRI-B). Med Oncol. 2013 Dec;30(4):743. doi: 10.1007/s12032-013-0743-0. Epub 2013 Oct 11. PMID 24114613